CLINICAL TRIAL: NCT06333574
Title: Clinical Randomized Controlled Trial of Weight Intervention to Improve Volumetric Load in Hemodialysis Patients
Brief Title: Weight Management of Dialysis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: qinxiu zhang (Other)
Responsible Party: Sponsor-Investigator, qinxiu zhang, Director, World Health Organization (WHO) Collaborating Centre, Chengdu University of Traditional Chinese Medicine
Organization: Chengdu University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDUTCM20240313
Record Dates: First submitted 2024-03-13; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Hemodialysis; Life Quality; Interdialytic Weight Gain; Cardiovascular Events; Hypertension; Dry Weight
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): received routine outpatient management. Specific methods: The dialysis doctor registered the information of the patient's weight and blood pressure at the end of dialysis, and informed the patient of the purpose, role and importance of weight management.
  Interventions: Other: Routine care
- Intervention group (Other): On the basis of routine outpatient management, patients or their family members were subjected to remote follow-up management based on wechat, and the follow-up time was 6 months. Specific methods: Same as the control group, the information of weight and blood pressure of the patients was registered at the end of dialysis, and the purpose, role and importance of weight management were informed to the patients. On this basis, a special wechat signal is set up to add patients or patients' family members as wechat friends and establish a wechat interaction platform with patients. In the interdialysis period, remind patients to weigh themselves through wechat (the time of each weighing is fixed, preferably consistent with the time of weighing in the hemodialysis center), control the weight gain during the interdialysis period not to exceed 4.5% of dry weight, and inform patients again about the purpose, role and importance of weight management.
  Interventions: Other: Family weight self-measurement and remote follow-up management based on wechat.

INTERVENTIONS:
Other: Family weight self-measurement and remote follow-up management based on wechat. — On the basis of routine outpatient management, patients or their family members were subjected to remote follow-up management based on wechat, and the follow-up time was 6 months. Specific methods: Same as the control group, the information of weight and blood pressure of the patients was registered at the end of dialysis, and the purpose, role and importance of weight management were informed to the patients. On this basis, a special wechat signal is set up to add patients or patients' family members as wechat friends and establish a wechat interaction platform with patients. In the interdialysis period, remind patients to weigh themselves through wechat (the time of each weighing is fixed, preferably consistent with the time of weighing in the hemodialysis center), control the weight gain during the interdialysis period not to exceed 4.5% of dry weight, and inform patients again about the purpose, role and importance of weight management.
  Arms: Intervention group
Other: Routine care — The dialysis doctor registered the information of the patient's weight and blood pressure at the end of dialysis, and informed the patient of the purpose, role and importance of weight management.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to Improve the quality of life in Hemodialysis patient. The main questions it aims to answer are:

* [Improve the self-compliance of dialysis patients with weight management]
* [alleviate the volume load of dialysis patients and reduce cardiovascular complications] Participants will be divided into two groups based on a weight management regimen： Control group: received routine outpatient management. Specific methods: The dialysis doctor registered the information of the patient's weight and blood pressure at the end of dialysis, and informed the patient of the purpose, role and importance of weight management.

Intervention group: On the basis of routine outpatient management, patients or their family members were subjected to remote follow-up management based on wechat, and the follow-up time was 6 months. Specific methods: Same as the control group, the information of weight and blood pressure of the patients was registered at the end of dialysis, and the purpose, role and importance of weight management were informed to the patients. On this basis, a special wechat signal is set up to add patients or patients' family members as wechat friends and establish a wechat interaction platform with patients. In the interdialysis period, remind patients to weigh themselves through wechat (the time of each weighing is fixed, preferably consistent with the time of weighing in the hemodialysis center), control the weight gain during the interdialysis period not to exceed 4.5% of dry weight, and inform patients again about the purpose, role and importance of weight management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18;
* Dialysis age ≥3 months;
* Survival ≥12 months;
* Patients themselves or family members can use wechat;
* Informed consent

Exclusion Criteria:

* Have a cognitive or intellectual disability unable to read and understand SMS;
* Have mental illness;
* Other serious complications occurred

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse event rate | 4, 8, and 12 weeks after intervention
  incidence of cardiovascular events (or hospitalization rate due to cardiovascular events such as hypertension and heart failure)
Rate of completion | 4, 8, and 12 weeks after intervention
  Completion rate of home self-measured weight combined with wechat intervention(including completion rate of home self-measured weight, completion rate of wechat intervention, and combination completion rate）

SECONDARY OUTCOMES:
dialysis related symptoms | 4, 8, and 12 weeks after treatment
  (fatigue, weakness, pruritus, dialysis patient quality of Life scale)
Laboratory index | 4, 8, and 12 weeks after treatment
  hemoglobin
level of Ga | 4, 8, and 12 weeks after treatment
  Laboratory index
level of P | 4, 8, and 12 weeks after treatment
level of PTH | 4, 8, and 12 weeks after treatment
level of K | 4, 8, and 12 weeks after treatment
level of Na | 4, 8, and 12 weeks after treatment
level of Cl | 4, 8, and 12 weeks after treatment
concentration of albumin and prealbumin | 4, 8, and 12 weeks after treatment
Laboratory index of total protein | 4, 8, and 12 weeks after treatment
Dialysis efficiency \ dialysis adequacy (KTV) | 4, 8, and 12 weeks after treatment
  Dialysis efficiency \ dialysis adequacy (KTV)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Yan B, Zhang S, Zhou Y, Zhang Q, Li X. Management of volume load for patients undergoing hemodialysis via WeChat and home monitoring in China: a protocol for a cluster-randomized trial. BMC Nephrol. 2025 Feb 6;26(1):58. doi: 10.1186/s12882-024-03932-0. PMID 39910544